CLINICAL TRIAL: NCT04470414
Title: COVID-19 IgG Antibodies in the Serum of Recovered Patients: a Longitudinal Study
Brief Title: COVID-19 IgG Antibodies in the Serum of Recovered Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam T. Amin, Assistant Lecturer, Assiut University
Other Study IDs: Cov-PH2020
Record Dates: First submitted 2020-07-12; First posted 2020-07-14 (Actual); Last update posted 2020-07-16 (Actual); Status verified 2020-07

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Recovered COVID-19 patients: Patients recovered from COVID-19 infection within three months before the start of the study.
  Interventions: Diagnostic Test: IgG antibodies immunoassay

INTERVENTIONS:
Diagnostic Test: IgG antibodies immunoassay — Assessment of IgG level will be done by quantitative assessment of IgG in the serum of recovered persons by Chemiluminescence Immunoassay (CLIA).

SUMMARY:
Coronavirus disease 2019 (COVID-19) is an infectious disease caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), which first appeared in China, in December 2019 and is now spreading worldwide and poses a great threat to public health. In 12th July 2020, the total number of cases worldwide was about 13 million cases with case fatality rate of 4.4% and in Egypt the total cases was 81158 and case fatality rate was 4.6%. (1,2).

In recent years, novel coronaviruses emerge periodically in different areas around the world. Severe acute respiratory syndrome coronavirus (SARS-CoV) occurred in 2002, which reportedly infected 8422 people with about 10% case fatality rate (3). Middle East respiratory syndrome coronavirus (MERS-CoV) was first identified in 2012 in Saudi Arabia, bringing a total of 1401 MERS-CoV infections, and about 35% case fatality rate (1). All the infection cases and recent epidemics show that coronaviruses impose a continuous threat to human beings and the economy as they emerge unexpectedly, spread easily, and lead to catastrophic consequences.

As the number of recovered patients with COVID-19 continues to be increasing, the strength and duration of immunity after infection is an important point to be studied. Moreover, understanding this issue is a critical point for controlling this epidemic as they are the key for herd immunity and for informing decisions on how and when to ease physical distancing restrictions and to be ready for other waves of the infection. There is currently no evidence if the people who have recovered from COVID-19 have antibodies and protected from a second attack of infection or future wave of this pandemic or not. Therefore, we will carry out a longitudinal study of immunity in recovered patients to assess SARS-Cov2 patients' risk for future reinfection.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥ 20 years.
* Prior COVID-19 infection confirmed by PCR detection of SARS-CoV-2 RNA or antigen in nasopharyngeal swab.
* Recovery from infection either confirmed by two consecutive negative PCR (collected ≥24 hours apart) or passing of 14 days since onset of COVID-19 symptoms and at least 3 days since resolution of fever without the use of antipyretics and improvement of respiratory symptoms

Exclusion Criteria:

* Presence of any chronic illness interfere with immunity (autoimmune diseases).
* Pregnancy.
* Recovery from three months or more.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients recovered from COVID-19 infection within three months before the start of the study.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Levels of IgG in the serum of recovered COVID-19 patients | 3rd, 6th and 12th months post infection
  Levels of IgG in the serum of recovered COVID-19 patients at different points during the first year of infection.

SECONDARY OUTCOMES:
Factors related to IgG level | 1 year
  The relationship between the IgG levels and severity of the disease, age of recovered patients and duration of symptoms and viral clearance.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud A. Abd El Aty, Prof., Study Director — Assiut University- Faculty of Medicine; Mariam T. Amin, Principal Investigator — Assiut University- Faculty of Medicine
Locations (1):
- Faculty of medicine- Assiut university, Asyut, Egypt

REFERENCES:
- [Background] Li G, Fan Y, Lai Y, Han T, Li Z, Zhou P, Pan P, Wang W, Hu D, Liu X, Zhang Q, Wu J. Coronavirus infections and immune responses. J Med Virol. 2020 Apr;92(4):424-432. doi: 10.1002/jmv.25685. Epub 2020 Feb 7. PMID 31981224
- [Background] Singhal T. A Review of Coronavirus Disease-2019 (COVID-19). Indian J Pediatr. 2020 Apr;87(4):281-286. doi: 10.1007/s12098-020-03263-6. Epub 2020 Mar 13. PMID 32166607
- [Background] Long QX, Tang XJ, Shi QL, Li Q, Deng HJ, Yuan J, Hu JL, Xu W, Zhang Y, Lv FJ, Su K, Zhang F, Gong J, Wu B, Liu XM, Li JJ, Qiu JF, Chen J, Huang AL. Clinical and immunological assessment of asymptomatic SARS-CoV-2 infections. Nat Med. 2020 Aug;26(8):1200-1204. doi: 10.1038/s41591-020-0965-6. Epub 2020 Jun 18. PMID 32555424
- See also: Coronavirus: Events as they happen — https://www.who.int/emergencies/diseases/novel-coronavirus-2019/events-as-they-happen
- See also: Coronavirus Update (Live): Cases and Deaths from COVID-19 Virus Pandemic — https://www.worldometers.info/coronavirus/